CLINICAL TRIAL: NCT00265434
Title: Nasal Inhalation of Dornase Alfa (Pulmozyme) in Patients With Cystic Fibrosis and Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: PD Dr. Joachim Riethmöller, Tübingen (Unknown); PD Dr. Assen Koitschev, Tübingen (Unknown); Dr. Gerlind Schneider (Unknown)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, Head of CF Center, Pediatric Pulmonology, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pilot-pulmozyme-nasal-cf
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis; Chronic Rhinosinusitis
MeSH Terms: conditions — Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dornase alfa (Active Comparator): DBPC-cross over trial
  Interventions: Drug: Pulmozyme
- isotonic saline (Placebo Comparator)
  Interventions: Drug: Pulmozyme

INTERVENTIONS:
Drug: Pulmozyme

SUMMARY:
Rhinosinusitis disorders are often associated with Cystic Fibrosis. They can restrict quality of life enormously and give cause to repeated ENT surgery. The basic defect in CF is a dysfunction of Chloride channels in exocrine glands, leading to retention of secretions and consecutive chronic inflammation with bacterial superinfections.

The prospective placebo controlled cross-over study aims at the evaluation of the efficacy of a nasally inhalation of Pulmozyme with respect to mucus retention and resulting inflammation.

ELIGIBILITY:
Inclusion Criteria (most important):

* Subject has a confirmed diagnosis of cystic fibrosis.
* Subject has chronic or recurrent rhinosinusitic disorders.
* Subject is 5 years or older.

Exclusion Criteria (most important):

* Subject has a critical condition (FEV1<30% and SaO2<93%).
* Subject had an ENT surgery within 6 months prior to study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Changes in sinonasal symptoms (SNOT-20 | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Jochen G. Mainz, M.D., Study Chair — University of Jena
Locations (1):
- Friedrich-Schiller-Universität, Jena, Thuringia, Germany

REFERENCES:
- [Background] Mainz JG, Schiller I, Ritschel C, Mentzel HJ, Riethmuller J, Koitschev A, Schneider G, Beck JF, Wiedemann B. Sinonasal inhalation of dornase alfa in CF: A double-blind placebo-controlled cross-over pilot trial. Auris Nasus Larynx. 2011 Apr;38(2):220-7. doi: 10.1016/j.anl.2010.09.001. Epub 2010 Oct 27. PMID 21030168